CLINICAL TRIAL: NCT03668990
Title: Feasibility, Validity and Reliability Kinematic Movement Analysis of Upper Limb Movements in Stroke and MS Patients Using Inertial Sensors
Brief Title: Feasability, Validty and Reliability of Inertial Sensors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: Revalidatie & MS Centrum Overpelt (Other); Jessa Hospital (Other)
Responsible Party: Principal Investigator, Peter Feys, Principal Investigator, Hasselt University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Kinematic01
Record Dates: First submitted 2017-09-14; First posted 2018-09-13 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Multiple Sclerosis; CVA
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- persons with Multiple Sclerosis (MS) (Other): 25 persons with MS Persons perform funtional-oriented upper limb movments while wearing IMUs (Xsens, MVN Studio). This is a full-body human measurement system based on inertial sensors, biomechanical models and sensor fusion algorithms applied in neurological patients for measuring upper limb movements.
  Funcitonal-oriented upper limb movements are performed at two different test days.
  Interventions: Other: IMUs (Xsens, MVN Studio)
- stroke patients (Other): 25 stroke patients Persons perform funtional-oriented upper limb movments while wearing IMUs (Xsens, MVN Studio). This is a full-body human measurement system based on inertial sensors, biomechanical models and sensor fusion algorithms applied in neurological patients for measuring upper limb movements.
  Funcitonal-oriented upper limb movements are performed at two different test days.
  Interventions: Other: IMUs (Xsens, MVN Studio)
- Healthy controls (Other): 50 healthy controls Persons perform funtional-oriented upper limb movments while wearing IMUs (Xsens, MVN Studio). This is a full-body human measurement system based on inertial sensors, biomechanical models and sensor fusion algorithms applied in neurological patients for measuring upper limb movements.
  Funcitonal-oriented upper limb movements are performed at two different test days.
  Interventions: Other: IMUs (Xsens, MVN Studio)

INTERVENTIONS:
Other: IMUs (Xsens, MVN Studio) — It is a full-body human measurement system based on inertial sensors, biomechanical models and sensor fusion algorithms applied in neurological patients for measuring upper limb movements.

SUMMARY:
This study has 3 aimes:

1. To investigate the feasibility of using IMUs (Xsens, MVN Studio) during functional tasks to assess upper limb kinematics in pwMS and stroke survivors. On the one hand, the feasibility of performing the tasks will be investigated . On the other hand, does the XSens give valuable data?
2. To investigate the discriminative validity of kinematic measurements of upper limb movements post-stroke and pwMS in comparison with gender and age-matched healthy controls
3. To investigate the test-retest reliability of the kinematic parameters collected during the different functional tasks in pwMS and stroke survivors

It is a cross-sectional case-controlled observational study, with 3 different groups: 25 Persons with Multiple sclerosis, 25 stroke patients and 50 healthy controls, matched by age and gender.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for all participants: Healthy controls, pwsMS and stroke patients

* No orthopedic or neuro-muscular impairments in the upper limb
* Age > 18 years
* Able to understand and execute the test instructions
* Perceived pain in one of the upper limbs of more than 4/10 (Visual Analog Scale)
* Able to move a joint (wrist, elbow or shoulder) in the upper limb against gravity without resistance (Medical Research Council) (16).

Inclusion criteria for PwMS:

- Diagnosed with MS using McDonald criteria (17)

Inclusion criteria Stroke patients

* First- ever single, unilateral (ischemic or hemorrhagic)
* At least one month after stroke
* No apraxia or hemi spatial neglect

Exclusion Criteria:

Exclusion Criteria for pwMS only:

* a relapse 3 months before the start of the study
* A change of symptomatic medication during the testing period

Exclusion Criteria:

- People with predominantly ataxia or tremor are excluded from the reliability part of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
kinematic parameter | day 2
  The data received of the IMU's are the angles of point task achievement (PTA). PTA is defined as the instant when the ROM, needed for successful task execution, was achieved. Different joint angles of PTA will be calculated by MVN BIOMECH software. Matlab (software version R2016b) and excel will be used to process the data.
kinematic parameter | day 3
  The data received of the IMU's are the angles of point task achievement (PTA). PTA is defined as the instant when the ROM, needed for successful task execution, was achieved. Different joint angles of PTA will be calculated by MVN BIOMECH software. Matlab (software version R2016b) and excel will be used to process the data.

SECONDARY OUTCOMES:
The Brunnström Fugl Meyer (BFM) | day 1
  The Brunnström Fugl Meyer (BFM) was used to measure motor control at the body functions and structures level. The upper limb section is applied: shoulder, elbow, forearm, wrist movements and grip
Action Research arm test | Day 1
  which assessed the patient's ability to handle objects varying in size
Trunk Impairment Scale | day 1
  To examine the clinimetric characteristics of the Trunk Impairment Scale (TIS). This scale evaluates motor impairment of the trunk after stroke. The TIS scores, on a range from 0 to 23, static and dynamic sitting balance as well as trunk co-ordination. It also aims to score the quality of trunk movement and to be a guide for treatment.
Manual Ability Measure-36 (questionnaire) | day1
  Perceived performance on activity level

CONTACTS AND LOCATIONS:
Overall Officials: peter Feys, prof. dr., Principal Investigator — Hasselt University; Joke Raats, drs, Study Chair — Hasselt University; Liesbet De Baets, dr., Study Chair — Hasselt University
Locations (2):
- Belgium (2):
  - Jessa Ziekenhuis, Hasselt
  - Revalidatie & MS Centrum Overpelt, Overpelt

IPD SHARING:
Plan to Share IPD: Undecided